CLINICAL TRIAL: NCT02073435
Title: A2ALL-Patients Safety System Improvements in Living Donor Liver Transplant
Brief Title: A2ALL-Patients Safety System Improvements in Living Donor Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Daniela Ladner, Assistant Professor, Northwestern University
Other Study IDs: A2ALL Safety Study; R01DK090129 (NIH)
Record Dates: First submitted 2013-06-20; First posted 2014-02-27 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Liver Diseases; Hepatocellular Cancer; Endstage Liver Disease; Liver Cirrhosis
Keywords: liver transplantation; living donor; Safety
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Post-Implementation Group: Living Donor Liver Transplant patients with evidence based donor pain management solution.
  Interventions: Behavioral: Donor pain management
- Pre-Implementation Group: Living Donor Liver Transplant patients prior to the implementation of the evidence based donor pain management solution.

INTERVENTIONS:
Behavioral: Donor pain management — The evidence-based donor pain management solution entails the following elements:
  Preoperative Assessment and Management:
  * Assessment of Patient Risk factors for Respiratory Depression (e.g. OSA Assessment: STOP BANG Questionnaire)
  * Bowel preparation (e.g. Colace or Golytely)
  * Patient Postoperative Pain Education - Educational handout on postoperative pain
  At the end of the case in OR:
  * Local Anesthetic (TAP block, OnQ device, intrathecal, local infiltration)
  * I.V. Ketorolac (when adequate hemostasis is determined by surgeon and urine output is > 500cc)
  * I.V. Steroids (Dexamethasone or Solumedrol)
  Postoperative Management:
  * NSAIDS x 72 hours followed by po cox-inhibitor until discharge (e.g. Celecoxib)
  * Opioids (Dilaudid PCA followed by oral opioids (e.g., Tylenol #3))
  Postoperative Assessment:
  o CO2 monitoring in PACU/ICU for early monitoring of respiratory depression
  Groups: Post-Implementation Group

SUMMARY:
Living donor liver transplantation (LDLT), involves complex systems and processes of care that are particularly vulnerable to medical errors and preventable complications. This ancillary study of the Adult-to-Adult Living Liver Transplantation Cohort Study (A2ALL) will focus on conducting a proactive, systematic, and comprehensive assessment of the vulnerabilities in the systems and process of LDLT care to reduce medical errors and preventable complications thereby improving the safety of LDLT care. This project will address an important gap in the knowledge needed to achieve high quality and safe LDLT care of patients by developing a process to: 1) proactively, systematically and comprehensively identify areas of vulnerabilities in LDLT care that can result in medical errors, 2) design and implement solutions to mitigate these weaknesses, and 3) evaluate the effectiveness of these solutions to improve the safety of LDLT care by measuring clinical and process outcomes before and after solution implementation across four A2ALL participating transplant centers

DETAILED DESCRIPTION:
This is an observational as well as a time-controlled study to be conducted at four participating A2ALL Deux Transplant Centers (TCs). The study is divided into three phases: an observational phase (Aim 1) to conduct a comprehensive and proactive patient safety risk assessment to describe preventable complications, near miss events, medical errors and hazardous conditions and in the delivery of standard of care to living donor liver transplant (LDLT) donors and recipients from the time of admission for the LDLT surgery through discharge after LDLT surgery. The in depth observational phase continues throughout the study and is scheduled to be completed by the end of the study (May 2015).

In phase 2-solution development and implementation phase (Aim 2): two high priority areas of care were identified for in depth assessment and solution development. The selection of the two high priority areas of LDLT standard of care was guided by the identification of vulnerabilities in the systems and processes of care with a high incidence and severity of related preventable complications and medical errors across the four participating A2ALL Deux TCs. To date, multiple priority areas were identified, based on the ongoing review of medical records (e.g., transition of care, glucose control, donor pain management, preoperative OR set-up). The participating A2ALL Deux TCs agreed to focus on an in depth assessment of the two areas that demonstrated high incidence and high severity of preventable complications and medical errors: 1) donor pain management and 2) preoperative OR set-up process.

1. Donor Pain Management:

   Upon further investigation, it was identified that living liver donors experience significant amount of pain, in the early postoperative period but also especially a few days after donation. Data from the four participating A2ALL Deux TCs reveal a 20% incidence, overall, of respiratory complications (e.g. re-intubation, requirement for application of Naloxone, etc.) directly related to the opioid use in the present LDLT standard of care for donor pain management. Based on these data, clinicians at the four participating A2ALL Deux TCs, in consultation with an international pain expert with particular expertise in transplantation (Paul White, MD University of Texas Southwestern Medical Center at Dallas, Dallas, Texas), developed an evidence-based donor pain management solution with the aim of reducing preventable complications as well as improving the donor pain experience. This evidence-based donor pain management solution was developed over months through in-person and telephone meetings of transplant surgeons, hepatologists, anesthesiologists and acute pain specialists from all four participating A2ALL Deux TCs, in addition to the research teams. Consensus has been reached on the key elements of the evidence-based donor pain management solution and all four participating A2ALL Deux TCs are poised to begin implementation.
2. Preoperative OR Set-up Process:

Preventable complications, near miss events, medical errors and hazardous conditions related to the preoperative OR set-up processes were identified. The four participating A2ALL Deux TCs will need to engage in additional review of the detailed assessment of the standardization and optimization of the preoperative OR set-up process and then, will collaboratively design a standardized process over a four month period (expected conclusion mid February 2014 in order to incorporate what occurs at the Collaborative at each site and overall). Solutions will be designed collaboratively to reduce the incidence and severity of related medical errors and preventable complications together with the TCs and their staff.

The measurement of solution impact to reduce preventable complications and medical errors (Aim 3) involves the implementation of the two collaboratively developed solutions: (1) Evidence-based donor pain management solution and (2) Standardization and optimization of the preoperative OR set-up process. During this phase relevant metrics pre- and post-implementation will be compared to assess the effectiveness of the implemented solutions.

ELIGIBILITY:
Inclusion Criteria:

A. Clinicians

1. Clinicians of both genders, of any race/ethnicity are included. Only clinicians who are unwilling to participate will be excluded.
2. Clinicians and staff who are involved in the care of LDLT donors and recipients (e.g., nurses, surgeons, anesthesiologists, hepatologists, unit secretaries from medical and surgical units, ICU, transplant coordinators, pharmacists) at the four participating A2ALL Deux TCs.

B. Patients

1. Every donor (≥ 21 years) and recipient involved in LDLT at the four participating A2ALL Deux TCs between 2004-2015, who were enrolled into the A2ALL cohort study Un and/or Deux. (However, to date medical record reviews were only performed for patients involved in LDLTs 2008 or later. Observations were initiated in December, 2011). After enrollment of patients into the A2ALL Deux cohort study ends (anticipated May 2014), all LDLT donors and recipients at the four participating A2ALL Deux TCs will be approached for enrollment into this ancillary A2ALL R01 patient safety study.
2. Patients have not been and will not be excluded on the basis of race, gender, or any other related characteristics.

Exclusion Criteria:

* No participants will be under 21 years of age. Patients will not be excluded on the basis of age, race, gender or any other non-employment related characteristics

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: CLINICIANS: All clinicians who are involved in the inpatient care provided to the LDLT A2ALL donors and recipients are eligible for the study. The group of clinicians eligible for the study involve all clinicians participating in the LDLT care between day of surgery through discharge: OR personnel (nurses, technicians, anesthesiologists, surgeons, research staff, cell saver staff, etc.), PACU/Intensive Care Unit personnel (nurses, anesthesiologists, surgeons, pharmacists, etc.) and floor personnel (nursing, coordinators, pharmacists, etc.).
  PATIENTS: Living Donor Liver Transplant patients (donor and recipients) from 2008-2015.
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ladner, MD MPH, Principal Investigator — Northwestern Univesity; Donna Woods, PhD, Principal Investigator — Northwestern University; Averell Sherker, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Lahey Clinic, Burlington, Massachusetts
  - Columbia University, New York, New York
  - Virginia Commonweath University-Medical College of Virginia, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Post-Implementation Group | Pre-Implementation Group
Started | 81 | 96
Completed | 81 | 96
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Post-Implementation Group | Pre-Implementation Group | Total
Number analyzed (Participants) | 81 | 96 | 177
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.96 (10.82) | 38.81 (11.04) | 38.88 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 81
  Male | 40 | 56 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 10 | 24
  Not Hispanic or Latino | 67 | 86 | 153
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 10 | 13
  White | 60 | 74 | 134
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Living Donor Pain Management
Description: Comparison of Average Pain Scores on Visual Analogue Pain Scale (0-10) measured before and after implementation of evidence-based donor pain management solution. 0 representing "No Pain", up through 10 representing "Worst possible, unbearable, excruciating pain".
Time Frame: Daily Visual Analogue Pain Scores (0-10) At transplant (post-operative day 0) and throughout hospitalization (post-operative days 1-8)
Measure: Mean (Standard Deviation); unit: Scores on Visual Analogue Pain Scale
Arm/Group | Post-Implementation Group | Pre-Implementation Group
Number analyzed (Participants) | 81 | 96
Scores on Visual Analogue Pain Scale
  Post-Operative Day 0 (Surgery Day) | 2.62 (1.85) | 2.56 (2.17)
  Post-Operative Day 1 | 2.87 (1.76) | 2.67 (1.42)
  Post-Operative Day 2 | 3.25 (1.89) | 2.79 (1.65)
  Post-Operative Day 3 | 3.56 (1.94) | 2.84 (1.93)
  Post-Operative Day 4 | 3.56 (1.90) | 3.14 (2.00)
  Post-Operative Day 5 | 3.11 (2.20) | 3.36 (2.14)
  Post-Operative Day 6 | 3.39 (2.04) | 4.10 (2.39)
  Post-Operative Day 7 | 3.47 (2.18) | 2.69 (2.18)
  Post-Operative Day 8 | 4.06 (2.92) | 2.81 (2.00)

2. Primary Outcome: Complications
Description: Cardiopulmonary complications
Time Frame: Perioperatively
Measure: Number; unit: Cardiopulmonary complications
Arm/Group | Post-Implementation Group | Pre-Implementation Group
Number analyzed (Participants) | 81 | 96
Cardiopulmonary complications | 0 | 12

ADVERSE EVENTS:
Description: When this study was originally created, it was designed as an interventional study with planned adverse event collection for those events that were related to study interventions. The study designed was then revised to observational only, and therefore adverse events were not collected since there were no longer study interventions.
Arm/Group | Post-Implementation Group | Pre-Implementation Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was originally intended to be a clinical trial, with control and intervention sites, however, per discussions with the NIDDK program officer the study design was changed to a observational study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No